CLINICAL TRIAL: NCT06569147
Title: A Phase I/II, Open Label, Study to Evaluate Safety, Tolerability and Efficacy of Elranatamab in Patients with Relapsed or Refractory AL Amyloidosis
Brief Title: Elranatamab in Patients with Relapsed or Refractory AL Amyloidosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Giada Bianchi, MD, Assistant Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-290
Record Dates: First submitted 2024-08-16; First posted 2024-08-23 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elranatamab Dose Schedule (Experimental): Phase I: Phase I will enroll up to 20 participants. All participants in Phase I will be hospitalized during Cycle 1 dosing. The first 5 participants will be hospitalized for 9 days, and subsequent participants will be hospitalized for 5 days. Elranatamab will be administered subcutaneously at a dose of 12 mg on C1D1, 32 mg on C1D4, and 76 mg on C1D8. Subsequent treatment doses will be 76 mg thereafter. If two or more participants at Level 0 experience DLT, dose will be decreased to Level -1. If 2 or more participants at Level -1 experience DLT, the trial will be discontinued.
  Phase II: All participants in Phase 2 will receive the RP2D determined in Phase 1. Phase 2 will enroll an additional 29 participants. If RP2D is determined to be Dose Level 0, the treatment schedule will be the same as described in Dose Level 0. If RP2D is determined to be Dose Level -1, the treatment schedule will be the same as described in Dose Level -1.Treatment duration is 6 cycles of 28 days per cycle.
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — Elranatamab administered subcutaneously for 6 cycles of treatment with 28 days in a treatment cycle
  Other Names: Elrexfio

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of elranatamab in patients with relapsed or refractory AL amyloidosis.

DETAILED DESCRIPTION:
This is a Phase I/II, multi-center, open-label study designed to evaluate the safety, tolerability and efficacy of elranatamab in patients with relapsed or refractory light chain (AL) amyloidosis. Phase 1 will enroll 4-20 participants, beginning enrollment at Dose Level 0. If two or more participants at Level 0 experience DLT, dose will be decreased to Level -1. Each participant will complete the 28-day dose-limiting toxicity (DLT) evaluation period prior to dosing the next patient. Assuming a recommended phase 2 dose (RP2D) is found, Phase 2 will enroll an additional 29 participants for a total of 49 participants.

Dose level 0 consists of: Cycle 1: 12 mg (D1)/32 mg (D4)/ 76 mg (D8, 15, 22); Cycle 2: 76 mg on D1, D8, D15 and D22. If < VGPR after Cycle 2: Cycles 3-6: 76 mg on D1, 8, 15 and 22. If ≥ VGPR after Cycle 2: Cycles 3-6: 76 mg on D1 and 15

Dose Level -1 consists of: Cycle 1: 12 mg (D1)/32 mg (D4)/ 76 mg (D8, D22), Cycles 2-6: 76 mg D1 and D15

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with AL amyloidosis based on IMWG criteria who have relapsed or refractory disease after treatment with at least one prior line of therapy (minimum 2 cycles).
* Participants must have progression of light chain disease, defined as dFLC >20mg/L.
* For Phase 2 only, measurable hematologic disease, satisfying one of the following criteria: Difference between involved and uninvolved free light chain (FLC) over 40 mg/L; Abnormal level of FLC with an abnormal κ/λ ratio (except in participants with CKD stage 3 or higher where a rise of lambda FLC to an abnormal level and of at least 50% over the nadir with a normal κ/λ ratio is acceptable); A serum M spike measuring ≥ 0.5 g/dL
* Age ≥ 18 years
* ECOG performance status ≤2 or Karnofsky ≥60%
* Participants must meet the following organ and marrow function as defined below: Absolute leukocyte count ≥3,000/mcL , Absolute neutrophil count ≥1,000/mcL, Absolute platelet count ≥75,000/mcL , Direct bilirubin ≤1.5 × institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN, Creatinine: Calculated clearance ≥30 mL/min using Cockcault-Groft equation
* Participants who received belantamab mafodotin are eligible if discontinued due to intolerance or adverse event.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* AL Amyloidosis Cardiac stage I, II or IIIa disease based on the 2013 European Modification of the 2004 Standard Mayo Clinic Staging in participants with advanced cardiac involvement (Dispenzieri et al., 2004; Wechalekar et al., 2013).
* The effects of elranatamab on the developing human fetus are unknown. Based on the mechanism of action, elranatamab may cause fetal harm when administered to a pregnant woman and therefore should not be used during pregnancy. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and until 90 days since the last dose of elranatamab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 90 days after completion of elranatamab administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Willingness to undergo study procedures, including bone marrow biopsies as detailed in the schedule of events.
* Participants should have received prior treatment with Daratumumab + CyBorD.

Exclusion Criteria:

* Prior BCMA-targeting bispecific antibodies or BCMA-targeting CAR-T therapy.
* Participants refractory to belantamab mafodotin OR participants that have received belantamab as the immediate past line of therapy.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Participants who are receiving any other investigational agents for this condition.
* Participants with Stage IIIB Amyloidosis as defined by the 2004 Mayo Clinic Criteria (see above).
* History of allergic reactions to elranatamab.
* Participants with an active malignancy (including lymphoma) with the following exceptions: adequately treated basal cell carcinoma, squamous cell carcinoma, or in situ cervical cancer; adequately treated stage I cancer from which the patient is currently in remission and has been for over 2 years; low-risk prostate cancer with a Gleason score < 7 and prostate specific antigen < 10ng/mL; other localized, indolent and/or low risk cancer may be permitted
* Women who are pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or 4 months following discontinuation of elranatamab, whichever is longer. Pregnant women are excluded from this study because elranatamab is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with elranatamab, breastfeeding should be discontinued if the mother is treated with elranatamab.
* Have any other medical, social or psychological factors that could affect the participant's safety or ability to consent personally or comply with study procedures.
* Participants meeting criteria for active MM based on presence of CRAB criteria (a ratio of involved versus uninvolved FLC over 100 is allowed in the absence of CRAB criteria).
* Participants with active clinically significant autoimmune diseases.
* Participants seropositive for the human immunodeficiency virus (HIV).
* Severe, uncontrolled orthostatic hypotension resulting in syncopal/pre-syncopal events despite optimized medical management (e.g., midodrine, pyridostigmine) and in the absence of volume depletion.
* Plan for autologous stem cell transplant during the first 6 months of protocol therapy.
* History of acute coronary syndrome or uncontrolled ventricular arrhythmias within 3 months prior to screening.
* Evidence of LV systolic dysfunction as defined by LVEF is < 30% by echocardiogram at Screening per site cardiology interpretation.
* Presence of severe valvular stenosis (e.g., aortic or mitral stenosis with a valve area < 1.0 cm2) or severe congenital heart disease.
* Have history of sustained ventricular tachycardia or aborted ventricular fibrillation or a history of atrioventricular nodal or sinoatrial nodal dysfunction if a permanent pacemaker (PPM) or implantable cardioverter-defibrillator (ICD) is not placed.
* QT corrected by Fridericia (QTcF) is > 550 msec on Screening ECG unless they have a PPM/ICD implanted.
* Screening EKG showing acute myocardial ischemia or active conduction system abnormalities with the exception of any of the following: First degree atrioventricular block; Second degree atrioventricular block Type 1 (Mobitz Type 1/Wenckebach type); Right or left bundle branch block (e.g., Left Bundle Branch Block, Right Bundle Branch Block, Left Anterior Fascicular Block, or Left Posterior Fascicular Block); Atrial fibrillation with a controlled ventricular rate; Bifascicular block assessed as benign by the Investigator
* Major surgery that required general anesthesia within 4 weeks of randomization or is planning major surgery during the study.
* NYHA class IV symptoms or participants with acute decompensation of congestive heart failure.
* Transplant eligible participants who have not undergone transplant are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
To determine RP2D | up to 26 months
  The recommended phase 2 dose determined in phase 1
To evaluate objective response rate (ORR) | up to 60 months
  Defined as the proportion of patients with CR, VGPR, or PR, and will be provided as unconfirmed and confirmed ORR at the end of six cycles of treatment. Confirmed responses are those that persist on repeat imaging study at least 28 days after the initial documentation of response.

SECONDARY OUTCOMES:
To assess safety and tolerability of elranatamab in patients with relapse or refractory AL amyloidosis | up to 72 months
  Number of participants with treatment-related adverse events as assessed by CTCAE version 5.0
To assess best overall response (BOR) | up to 72 months
  BOR will be analyzed as the number of patients (percentage) with each response, divided by the number of patients treated.
To assess duration of response (DoR) | up to 72 months
  DoR will be analyzed using Kaplan-Meier method and is defined as the time from the first documentation of CR, VGPR, or PR to the first documentation of objective progression or death due to any cause. .
To assess progression-free survival (PFS) | up to 72 months
  Progression-free Survival (PFS) will be analyzed using Kaplan-Meier method and is defined as the time from Cycle 1 Day 1 to first documentation of objective progression (PD) or death due to any cause, whichever comes first.
To assess overall survival (OS) | up to 72 months
  OS is defined as the time from the date of Cycle 1 Day 1 to date of death due to any cause.
Incidence and severity of cytokine release syndrome (CRS) and immune effector cell- associated neurotoxicity syndrome (ICANS) | up to 72 months
  Number of cases of CRS and ICANs and Grade of CRS and ICANs cases
Incidence of treatment emergent adverse events | up to 72 months
  Number of treatment- emergent AEs. An AE is treatment-emergent if the onset occurs on Cycle 1 Day 1 through 90 days after the last dose of investigational product.
To assess major organ deterioration (MOD) progression free survival (PFS) for the duration of the study | up to 72 months
  PFS is defined as the time from Cycle 1 Day 1 to first documentation of objective progression (PD) or death due to any cause, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Giada Bianchi, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States